CLINICAL TRIAL: NCT05653180
Title: A Single Arm,Multi-center,Phase Ib/II Clinical Study Evaluating IBI310 Combined With Sintilimab in Patients With Advanced Biliary Tract Cance(BTC)
Brief Title: IBI310 in Combination With Sintilimab in Patients With Advanced Biliary Tract Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI310J201
Record Dates: First submitted 2022-12-06; First posted 2022-12-16 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Advanced Biliary Tract Cancer
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI310+ sintilimab (Experimental): All Subjects will be treated with : Sintilimab 200mg IV Q3W continuously and IBI310 2mg/kg IV single dose, 3 weeks later, IBI310 maintenance dose is 1mg/kg IV Q6W until progression (treatment duration up to 24 months).
  Interventions: Drug: IBI310; Drug: sintilimab

INTERVENTIONS:
Drug: IBI310 — 2mg/kg IV,3 weeks later, 1mg/kg IV Q6W
Drug: sintilimab — 200mg IV Q3W
  Other Names: IBI308

SUMMARY:
This research study is designed to establish whether the combination of IBI310 & Sintilimab has efficacy in patients with advanced BTC

ELIGIBILITY:
Inclusion Criteria:

1. The subject must sign the written informed consent form, and can comply with the visits and related procedures specified in the protocol.
2. Aged ≥18 years.
3. Patients with unresectable or relapsed or metastatic advanced Biliary tract cancer,and diagnosed by histology/cytology (except carcinoma of ampulla).
4. Had progressed after receiving at least first-line systemic treatment (if a patient has progressed within 6 months after receiving systemic treatment during adjuvant chemotherapy or concurrent radiochemotherapy, she will be deemed to have received first-line treatment).
5. Patients who have never received any anti-PD-1, anti-PD-L1/L2 antibody, anti-CTLA-4 antibody, or other immunotherapy.
6. The subject must have at least one measurable lesion as the target lesion (according to RECIST V1.1). A measurable lesion in the radiation field from previous radiotherapy or local treatment, can also be chosen as the target lesion if confirmed progression.

Exclusion Criteria:

1. Diagnosis of other malignant tumors within 5 years before the first administration, excluding radically cured skin basal cell carcinoma, skin squamous cell carcinoma, radically resected carcinoma in situ and/or thyroid papillary carcinoma.
2. Patients who have previously received organ or bone marrow transplantation.
3. Patients with acute or chronic active hepatitis B or C infection, hepatitis B virus (HBV) DNA> 2000 IU/ml or 104 copies/ml; hepatitis C virus (HCV) antibody positive and HCV-RNA >103 copies/ml;. Patients with acute or chronic active hepatitis B or C infection who have received nucleotide antiviral therapy and are below the above standards can be selected.
4. Uncontrollable hypertension, systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg after best medical treatment, history of hypertensive crisis or hypertensive encephalopathy.
5. Pleural effusion, ascites, and pericardial effusion with clinical symptoms or requiring drainage , patients who only shows with a few pleural effusion, ascites, and pericardial effusion by imaging and with no clinical symptoms can be selected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 24 months
  Investigator evaluated ORR per RECIST V1.1

SECONDARY OUTCOMES:
progression free survival, PFS | up to 24 months
  PFS is defined as the time from first treatment to the date of the first documented tumor progression as determined by the investigator (per RECIST 1.1), or death due to any cause.
duration of response, DoR | up to 24 months
  Defined as the time from the first documented objective response to the first documented progressive disease or death of any cause, whichever occurs first;
disease control rate, DCR | up to 24 months
  Defined as the proportion of patients whose best response is CR, PR, and stable disease (SD) non-CR/non-PD
Overall Survival,OS | up to 24 months
  OS is defined as the time from enrollment to the date of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan cancer Hospital, Changsha, Hunan, China